CLINICAL TRIAL: NCT01790971
Title: Low Dose Spinal Morphine for Patients With Obstructive Sleep Apnea (OSA) Undergoing Total Hip Arthroplasty (THA)
Brief Title: Spinal Morphine for Patients With Obstructive Sleep Apnea
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: competing studies
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-0460-A
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Spinal morphine
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal morphine (Active Comparator): 100μg of morphine will be added to the intrathecal mixture.
  Interventions: Drug: Intrathecal Morphine
- No Intrathecal morphine (Active Comparator): Morphine will not be added to the intrathecal mixture.
  Interventions: Drug: No Intrathecal Morphine

INTERVENTIONS:
Drug: Intrathecal Morphine — Depending on the randomization schedule, 100μg of morphine will or will not be added to the intrathecal mixture.
  Other Names: Kadian
  Arms: Intrathecal morphine
Drug: No Intrathecal Morphine — Depending on the randomization schedule, 100μg of morphine will or will not be added to the intrathecal mixture.
  Other Names: Kadian
  Arms: No Intrathecal morphine

SUMMARY:
Patients with Obstructive Sleep Apnea (OSA) appear to be especially vulnerable to medications that suppress pharyngeal muscle activity such as general anesthetics and opioids. Opioids can depress the ventilator response to airway obstruction and inhibit the awakening response to hypoxia and hypercarbia, resulting in central respiratory depression. OSA is therefore an important risk factor for serious postoperative complications, including perioperative death. While OSA is increasingly recognized as a serious perioperative concern, current clinical practices are highly inconsistent with regard to the management of surgical patients with OSA. Additionally, the relative safety of intrathecal opioids in this patient population remains unknown.

DETAILED DESCRIPTION:
Total hip and knee arthroplasty (THA and TKA) are among the most common orthopedic procedures performed worldwide1. They have been shown to reduce chronic pain, increase the ability to function independently, and improve quality of life2,3. With an aging and increasingly obese North American population, the uses of THA and TKA are increasing 4. One of the main challenges associated with THA as well as TKA continues to be the perioperative management of patients who are elderly or obese, and their associated co-morbidities. Both THA and TKA are commonly performed under neuraxial anesthesia. Neuraxial anesthesia has been reported to provide multiple benefits when compared to general anesthesia and/or systemic analgesia including superior post-operative analgesia5, reduced opioid consumption6, improved rehabilitation7, and reduced morbidity and mortality8-12. The addition of opioids to the neuraxial local anesthetic solution has been common practice since 1979, when morphine was first shown to provide effective and prolonged analgesia after intrathecal administration13. For both THA and TKA surgeries, intrathecal morphine provides effective analgesia14-16 allowing for a reduction of the dose of intrathecal local anesthetic (thus minimizing side effects)17, and has a marked postoperative opioid-sparing effect14-16. However, these benefits of intrathecal morphine must be weighed against its risks of pruritis, nausea/vomiting, urinary retention, and, of most concern, respiratory depression18.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, aged 18-85
2. ASA physical status I-III
3. Suspected of having Obstructive Sleep Apnea(OSA) or previously diagnosed with OSA
4. Scheduled to undergo elective primary Total Hip or Knee Arthroplasty

Exclusion Criteria:

1. Chronic obstructive pulmonary disease
2. Asthma
3. History of congestive heart failure
4. Valvular disease
5. Dilated cardiomyopathy
6. Implanted pacemaker or defibrillator
7. Diagnosed OSA who are undergoing continuous positive airway pressure (CPAP) treatment
8. Contraindications to spinal anesthesia
9. Contraindications to a component of multi-modal analgesia
10. Local anesthetic allergy
11. Anticipated surgical duration > 2.5hrs
12. Opioid tolerance (>250mg/24hr oral morphine equivalent pre-operatively)
13. Pregnancy
14. History of significant cognitive or psychiatric condition that may affect patient assessment, or
15. Inability to provide informed consent.
16. Participation in other clinical studies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Average Oxygen Desaturation Index (ODI) for the first 72 hours postoperatively. | 72 hours
  Oxygen Desaturation Index (ODI) is defined as the average number of episodes of desaturation ≥ 4% lasting at least 10 seconds, per hour of sleep. ODI will be measured with a nocturnal pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, Principal Investigator — University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Liu SS, Wu CL. The effect of analgesic technique on postoperative patient-reported outcomes including analgesia: a systematic review. Anesth Analg. 2007 Sep;105(3):789-808. doi: 10.1213/01.ane.0000278089.16848.1e. PMID 17717242